CLINICAL TRIAL: NCT00060372
Title: CTLA-4 Blockade With MDX-010 to Induce Graft-Versus-Malignancy Effects Following Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Ipilimumab After Allogeneic Stem Cell Transplant in Treating Patients With Persistent or Progressive Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00042; 040749; P-6082; NCI-6082; CDR0000301644; R01CA093891 (NIH)
Record Dates: First submitted 2003-05-06; First posted 2003-05-07 (Estimated); Last update posted 2013-03-27 (Estimated); Status verified 2013-03

CONDITIONS: Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Atypical Chronic Myeloid Leukemia, BCR-ABL1 Negative; Childhood Myelodysplastic Syndromes; Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Disseminated Neuroblastoma; Malignant Neoplasm; Ovarian Choriocarcinoma; Ovarian Embryonal Carcinoma; Ovarian Immature Teratoma; Ovarian Mature Teratoma; Ovarian Mixed Germ Cell Tumor; Ovarian Monodermal and Highly Specialized Teratoma; Ovarian Polyembryoma; Ovarian Yolk Sac Tumor; Previously Treated Myelodysplastic Syndromes; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Malignant Testicular Germ Cell Tumor; Recurrent Mantle Cell Lymphoma; Recurrent Neuroblastoma; Recurrent Ovarian Epithelial Cancer; Recurrent Ovarian Germ Cell Tumor; Refractory Chronic Lymphocytic Leukemia; Refractory Multiple Myeloma; Relapsing Chronic Myelogenous Leukemia; Stage I Multiple Myeloma; Stage II Multiple Myeloma; Stage II Ovarian Epithelial Cancer; Stage III Malignant Testicular Germ Cell Tumor; Stage III Multiple Myeloma; Stage III Ovarian Epithelial Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Stage IV Breast Cancer; Stage IV Ovarian Epithelial Cancer; Testicular Choriocarcinoma; Testicular Choriocarcinoma and Embryonal Carcinoma; Testicular Choriocarcinoma and Seminoma; Testicular Choriocarcinoma and Teratoma; Testicular Choriocarcinoma and Yolk Sac Tumor; Testicular Embryonal Carcinoma; Testicular Embryonal Carcinoma and Seminoma; Testicular Embryonal Carcinoma and Teratoma; Testicular Embryonal Carcinoma and Teratoma With Seminoma; Testicular Embryonal Carcinoma and Yolk Sac Tumor; Testicular Embryonal Carcinoma and Yolk Sac Tumor With Seminoma; Testicular Teratoma; Testicular Yolk Sac Tumor; Testicular Yolk Sac Tumor and Teratoma; Testicular Yolk Sac Tumor and Teratoma With Seminoma
MeSH Terms: conditions — Congenital Abnormalities; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Neoplasms; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Follicular; Testicular Neoplasms; Lymphoma, Mantle-Cell; Neuroblastoma; Carcinoma, Ovarian Epithelial; Leukemia, Lymphocytic, Chronic, B-Cell; Multiple Myeloma; Breast Neoplasms; Carcinoma, Embryonal; Seminoma; Teratoma; Endodermal Sinus Tumor; Teratoma, Testicular | interventions — Ipilimumab; CTLA-4 Antigen

ARMS (1):
- Treatment (ipilmumab and donor lymphocyte infusion) (Experimental): Patients receive ipilimumab IV over 90 minutes. Cohorts of 3-6 patients receive escalating doses of ipilimumab until the MTD is determined. The MTD is the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Patients with persistent or progressive disease at 60 days after ipilimumab administration and no evidence of graft-versus-host disease receive donor lymphocyte infusions every 60 days for a total of 3 infusions.
  Interventions: Drug: ipilimumab; Drug: therapeutic allogeneic lymphocytes

INTERVENTIONS:
Drug: ipilimumab — Given IV
  Other Names: anti-cytotoxic T-lymphocyte-associated antigen-4 monoclonal antibody; MDX-010; MDX-CTLA-4; monoclonal antibody CTLA-4
Drug: therapeutic allogeneic lymphocytes — Given IV
  Other Names: ALLOLYMPH

SUMMARY:
This phase I trial is studying how well ipilimumab works after allogeneic stem cell transplant in treating patients with persistent or progressive cancer. Monoclonal antibodies can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the dose of MDX-010 (ipilimumab) that can safely be administered to patients with persistent or progressive malignancy following allo-HCT.

II. To determine the pharmacokinetics of different doses of MDX-010 administered as a single dose to patients with persistent or progressive malignancy following allo-HCT.

III. By assessment of aims 1 and 2, to determine the best dosing regimen for further study of CTLA-4 blockade in conjunction with escalating dose donor-leukocyte infusions (DLI) in patients with evidence of residual or progressive malignancy following allo-HCT.

IV. To assess if there is preliminary evidence of efficacy following the administration of MDX-010 in this population.

OUTLINE:

Patients receive ipilimumab intravenously (IV) over 90 minutes.

Cohorts of 3-6 patients receive escalating doses of ipilimumab until the maximum tolerated dose (MTD) is determined. The MTD is the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients with persistent or progressive disease at 60 days after ipilimumab administration and no evidence of graft-versus-host disease receive donor lymphocyte infusions every 60 days for a total of 3 infusions.

Patients are followed at 4, 5, 6, 9, and 12 months and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of persistent or progressive hematologic malignancy or solid tumor after allogeneic hematopoietic stem cell transplantation (AHSCT)
* Patients are eligible for study entry at any time between post-transplantation day 90 and 3 years after withdrawal of immunosuppressive therapy
* Acute myeloid leukemia (AML) or acute lymphoblastic leukemia (ALL) that meets any of the following criteria: hematologic relapse by standard criteria, hematologic persistence evidenced by bone marrow blasts > 10% after day 30 post-AHSCT
* Cytogenetic progression as evidenced by an increase in the percentage of Philadelphia chromosome (Ph)1-positive metaphases (or Ph1-positive cells by fluorescent in situ hybridization) from complete cytogenetic response (0% Ph1-positive cells) to partial response (1-34% Ph1-positive cells); PR to minor response (35-94% Ph1-positive cells); or MR to no response (95-100% Ph1-positive cells)
* Resistance to imatinib mesylate, defined as disease progression (hematologic, cytogenetic, or molecular) during OR failure to respond to (i.e., lack of complete hematologic response after 3 months, lack of partial cytogenetic response after 6 months, or lack of complete cytogenetic response after 12 months) prior imatinib mesylate therapy
* Myelodysplastic syndromes that meet any of the following criteria:

Hematologic relapse by standard criteria, cytogenetic relapse evidenced by recurrence of clonal abnormality in patients who achieved CCR after AHSCT, hematologic persistence evidenced by cytopenias not attributable to other post-transplant causes accompanied by characteristic morphological changes more than 90 days after AHSCT

* OR; Hematologic persistence evidenced by cytopenias not attributable to other post-transplant causes accompanied by characteristic morphological changes more than 90 days after AHSCT, or cytogenetic persistence evidenced by persistence of clonal abnormality more than 90 days after AHSCT
* Chronic lymphocytic leukemia that meets any of the following criteria:

greater than 25% increase in absolute lymphocytosis of > 5,000/mm3, greater than 25% increase in measurable lymphadenopathy, persistence of absolute lymphocytosis of > 5,000/mm3 at day 90 or later after AHSCT, persistence of lymphadenopathy of ≥ 3 cm in diameter at day 90 or later after AHSCT

* Aggressive non-Hodgkin's lymphoma (e.g., diffuse large cell lymphoma, lymphoblastic lymphoma, mantle cell lymphoma, or peripheral T cell lymphoma), Hodgkin's lymphoma, OR solid tumor that meets any of the following criteria: greater than 50% increase in measurable or evaluable disease, persistence of measurable lesions > 3.0 cm in diameter at day 90 or later after AHSCT OR;
* Persistence of malignancy by biopsy or positron emission tomography scan unless there is clear evidence of progression
* Multiple myeloma with demonstrated resistance to or intolerance of prior thalidomide and bortezomib unless these agents are contraindicated (e.g., due to peripheral neuropathy) and meeting any of the following criteria: greater than 25% increase in paraprotein band, abnormal quantitative immunoglobulin level, or urine protein excretion OR
* Greater than 25% increase in percent of plasma cells in the bone marrow (if > 15%), presence of new lytic bone lesions, new extramedullary lesions OR ≥ 25% enlargement of existing extramedullary lesions, persistence of paraprotein band, abnormally elevated quantitative immunoglobulin level, or bone marrow plasmacytosis > 15% for a period of at least 90 days after AHSCT
* At least 1 bidimensionally measurable lesion ≥ 1.5 cm in diameter
* Evaluable disease is defined as disease that is assessable for response (e.g., pleural effusion, elevated serum tumor)
* Bone metastases that can be assessed by CT scan or MRI considered evaluable
* Leukemia is considered evaluable disease
* Patients who met criteria for persistence or progression with AML, ALL, CML, or aggressive NHL AND are currently in complete remission after reinduction therapy do not require measurable or evaluable disease to be eligible
* At least 50% donor chimerism in the T-cell lineage OR full (≥ 90%) donor chimerism in unseparated blood on last assessment within 3 months before study entry
* No evidence on consecutive testing of > 10% decline in T-cell chimerism beyond the error of the test
* ECOG 0-2
* Life expectancy: More than 3 months
* No prior grade 3 or 4 acute graft-vs-host disease
* No concurrent autoimmune diseases requiring the chronic use of immunosuppressive medications, active connective tissue disease, CNS disease including multiple sclerosis or demyelinating disease, inflammatory bowel disease, autoimmune hepatitis
* No ongoing serious infection
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 4 months after study therapy
* No other serious ongoing medical condition that would preclude study participation
* No other malignancy within the past 5 years
* No psychological or psychiatric condition that would preclude study participation
* No prior anti-cytotoxic T-lymphocyte-associated antigen-4 monoclonal antibody (MDX-010)
* At least 6 weeks since prior immunosuppressive agents
* At least 2 weeks since prior imatinib mesylate
* No concurrent imatinib mesylate
* At least 6 weeks since prior and no concurrent immunosuppressive agents for clinically active graft-versus-host disease (GVHD) prophylaxis or treatment
* No other concurrent investigational agents
* OR Cytogenetic persistence evidenced by any Ph1-positive metaphases in bone marrow after day 90 post-AHSCT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2003-04; Primary Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Incidence of grade 3 and 4 acute GVHD based on NCI CTC | 60 days following administration of ipilimumab
Incidence of graft rejection following ipilimumab defined as the percentage of patients entered who demonstrate =< 10% donor T-cell chimerism | Post-infusion day 60
Autoimmune reaction defined as >= grade 3 dysfunction of a vital organ or the graft | Up to 5 years

SECONDARY OUTCOMES:
Polyclonal T-cell activation monitored by clinical assessment and laboratory evidence (anti CD3, CD4, CD8) and markers of activation (anti CD69, CD25, CD44 and MHC class II) | Up to 5 years
Incidence of extensive stage chronic GVHD | Post-infusion day 360
Disease response | Up to day 360 post ipilimumab infusion
Disease-free survival | Up to day 360 following antibody infusion
  Kaplan- Meier estimates of probability will be used.
Overall survival | Up to 360 days post-infusion
  Kaplan- Meier estimates of probability will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Ewa Carrier, Principal Investigator — University of California, San Diego
Locations (5):
- United States (5):
  - Scripps Clinic - La Jolla, La Jolla, California
  - University of California San Diego, La Jolla, California
  - Blood and Marrow Transplant Group of Georgia, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Dana-Farber Harvard Cancer Center, Boston, Massachusetts

REFERENCES:
- [Derived] Bashey A, Medina B, Corringham S, Pasek M, Carrier E, Vrooman L, Lowy I, Solomon SR, Morris LE, Holland HK, Mason JR, Alyea EP, Soiffer RJ, Ball ED. CTLA4 blockade with ipilimumab to treat relapse of malignancy after allogeneic hematopoietic cell transplantation. Blood. 2009 Feb 12;113(7):1581-8. doi: 10.1182/blood-2008-07-168468. Epub 2008 Oct 30. PMID 18974373